CLINICAL TRIAL: NCT07185555
Title: Applying Very Low Calorie Ketogenic Diet to the Treatment of Obesity in People With Type 1 Diabetes on Intensive Insulin Therapy Using Automated Insulin Delivery System
Brief Title: Vey Low-Energy Ketogenic Therapy in Adults With Type 1 Diabetes and Obesity on Intensive Insulin Therapy Using Advanded Hybrid Closed Loop System
Acronym: KET1D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Principal Investigator, Francesco Giorgino, Professor of Endocrinology, Director of Department of Precision and Regenerative Medicine and Ionian Area, Chief of Division of Endocrinology - University Hospital Policlinico Consorziale, Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1835/CEL
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes (T1D); Obesity (Disorder)
Keywords: Type 1 Diabetes Mellitus; Obesity; Very Low-Energy Ketogenic Diet; Insulin Therapy; Weight Loss; Continuous Glucose Monitoring; Advanced Hybrid Closed Loop
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Very Low-Energy Ketogenic Therapy with Advanced Hybrid Closed Loop in Adults with T1D and Obesity (Experimental): Participants will undergo a 4-week Very Low-Energy Ketogenic Therapy (600-800 kcal/day) using commercial meal replacements with very low carbohydrate content, high biological value proteins (milk, whey, pea, soy), and added fiber (inulin, FOS). Gluten-free, lactose-free, and vegan options will be available. Therapy will be performed while continuing intensive insulin treatment with an Advanced Hybrid Closed Loop (AHCL) system. Participants will perform daily self-monitoring of capillary ketonemia, maintain hydration, and abstain from intense exercise. Follow-up visits at weeks 1, 2, 3, and 4 will assess safety, metabolic control, and weight loss. After completion, a structured reintroduction of conventional meals will be initiated.
  Interventions: Dietary Supplement: VLEKT

INTERVENTIONS:
Dietary Supplement: VLEKT — Participants will follow a Very Low-Energy Ketogenic Therapy (VLEKT) providing 600-800 kcal/day for 4 weeks. The intervention consists of meal replacements (solid or liquid, ready-to-use or reconstituted) with very low carbohydrate content, high-quality proteins (milk, whey, pea, soy), and fiber (inulin, FOS). Gluten-free, lactose-free, and vegan options are available. Meal replacements are provided by Therascience or Penta at discounted prices. Participants will self-monitor capillary ketonemia daily, maintain adequate hydration, and avoid intense physical exercise. The Advanced Hybrid Closed Loop (AHCL) insulin delivery system will be used throughout the study with periodic adjustments based on device downloads. At the end of the 4-week intervention, a structured reintroduction of conventional meals will be initiated.

SUMMARY:
Overweight and obesity are frequent in adults with type 1 diabetes (T1D), with prevalence exceeding 50% in recent studies. Excess weight in T1D is associated with higher cardiometabolic risk and therapeutic challenges, while effective and safe weight management strategies are still limited.

This single-center, single-arm feasibility study will evaluate the efficacy and safety of a Very Low-Energy Ketogenic Therapy (VLEKT; 600-800 kcal/day) in adults with T1D and obesity treated with Advanced Hybrid Closed Loop (AHCL) insulin delivery systems. Participants will follow a structured 4-week program with commercial very-low-carbohydrate, high-protein meal replacements, under close medical supervision.

The primary endpoint is change in body weight at 4 weeks. Secondary outcomes include body composition, muscle strength, glucose metrics, insulin requirements, biochemical parameters, and patient-reported outcomes. Safety will be assessed through hypoglycemia incidence, ketone monitoring, and occurrence of diabetic ketoacidosis (DKA).

The study will enroll 14 participants. It is expected that VLEKT will achieve ~5% weight loss within one month while maintaining glycemic safety under AHCL technology.

DETAILED DESCRIPTION:
Excess weight in type 1 diabetes (T1D) is increasingly recognized as a critical clinical problem. Factors contributing to weight gain include intensive insulin therapy, compensatory intake of high-energy foods to prevent hypoglycemia, reduced physical activity due to fear of hypoglycemia, and pathophysiological mechanisms such as adipose tissue dysfunction and insulin resistance. Current therapeutic options for weight management in T1D are limited compared with type 2 diabetes, and novel approaches are urgently needed.

Ketogenic and very low-carbohydrate diets are effective in obesity and type 2 diabetes but have traditionally been discouraged in T1D because of risks of hypoglycemia, dyslipidemia, poor adherence, and diabetic ketoacidosis (DKA). The introduction of Advanced Hybrid Closed Loop (AHCL) systems, which combine continuous glucose monitoring with automated insulin delivery, provides a safer framework to test structured dietary interventions that were previously considered unsuitable in this population.

This feasibility study investigates a Very Low-Energy Ketogenic Therapy (VLEKT) for 4 weeks in adults with T1D and obesity using AHCL technology. The intervention will consist of commercially available meal replacements (600-800 kcal/day, <30 g/day carbohydrates, adequate protein supply) with strict monitoring of capillary ketones and insulin adjustments.

Baseline assessments include anthropometry, bioimpedance-derived body composition, handgrip strength, biochemical testing, continuous glucose monitoring metrics, and validated questionnaires (SF-12, IPAQ, PSQI, FH-15). Participants will attend weekly visits for clinical review, adherence reinforcement, safety checks, and repeat assessments. At study completion, a gradual reintroduction of conventional meals will be initiated.

The primary endpoint is absolute weight change after 4 weeks. Secondary endpoints include proportion achieving ≥5% weight loss, changes in body composition and muscle strength, glucose control (TIR, TAR, TBR, CV, GMI, GRI, TITR), insulin requirements, lipid and liver function markers, and patient-reported outcomes. Safety evaluation will focus on hypoglycemia incidence and DKA events.

Sample size calculation determined that 14 participants are required to detect a clinically relevant mean weight reduction of ~5%. The results will provide initial evidence on the feasibility, metabolic impact, and safety of VLEKT in this specific population, laying the groundwork for larger randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

Diagnosis of type 1 diabetes or autoimmune diabetes for ≥ 12 months

BMI ≥ 30 kg/m²

HbA1c < 9%

Knowledge and use of carbohydrate counting

Use of an Advanced Hybrid Closed Loop (AHCL) system for ≥ 3 months and willingness to maintain it during the study

At least 1 diabetology follow-up visit in the last 12 months (including telemedicine)

Willingness to purchase meal replacements for the entire study duration

Exclusion Criteria:

Ketoacidosis, severe hypoglycemia with seizures/coma, or severe hyperglycemia requiring hospitalization in the last 6 months

Febrile illness within the last 2 weeks

Dietary restrictions or intolerances incompatible with study food supplies

Celiac disease, gastroparesis, food allergies

Intense physical exercise >2 hours on >3 days per week

History or risk of eating disorder, or other psychiatric disorders

Recreational drug use or excessive alcohol consumption

Chronic kidney disease (eGFR <60 ml/min)

Gallstones

Liver failure

Heart failure (NYHA III-IV), unstable angina, cardiac arrhythmia, myocardial infarction, or stroke within the last 12 months

Respiratory failure

Severe or active infections

Planned elective surgery

Rare metabolic diseases (porphyria, CPT2 deficiency, mitochondrial fatty acid oxidation defect, pyruvate carboxylase defect)

Pregnancy (current or actively trying to conceive)

Breastfeeding

Current glucocorticoid therapy (except stable low-dose, inhaled, or replacement for adrenal insufficiency)

Other serious medical conditions that might interfere with participation or study completion in the investigator's judgment

Participant judged unable or unwilling to complete the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2025-12-14 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in body weight from baseline to end of 4-week Very Low-Energy Ketogenic Therapy | Baseline and Week 4
  Body weight will be measured in kilograms using a calibrated scale at baseline and after completion of the 4-week intervention. The primary outcome is the absolute change in weight from baseline. Participants will be assessed under standardized conditions (light clothing, no shoes, fasting state where possible).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Policlinico Consorziale, Bari, Italy, Italy

REFERENCES:
- [Background] Barrea L, Caprio M, Grassi D, Cicero AFG, Bagnato C, Paolini B, Muscogiuri G. A New Nomenclature for the Very Low-Calorie Ketogenic Diet (VLCKD): Very Low-Energy Ketogenic Therapy (VLEKT). Ketodiets and Nutraceuticals Expert Panels: "KetoNut", Italian Society of Nutraceuticals (SINut) and the Italian Association of Dietetics and Clinical Nutrition (ADI). Curr Nutr Rep. 2024 Sep;13(3):552-556. doi: 10.1007/s13668-024-00560-w. Epub 2024 Jul 23. PMID 39039372
- [Background] Phillip M, Nimri R, Bergenstal RM, Barnard-Kelly K, Danne T, Hovorka R, Kovatchev BP, Messer LH, Parkin CG, Ambler-Osborn L, Amiel SA, Bally L, Beck RW, Biester S, Biester T, Blanchette JE, Bosi E, Boughton CK, Breton MD, Brown SA, Buckingham BA, Cai A, Carlson AL, Castle JR, Choudhary P, Close KL, Cobelli C, Criego AB, Davis E, de Beaufort C, de Bock MI, DeSalvo DJ, DeVries JH, Dovc K, Doyle FJ, Ekhlaspour L, Shvalb NF, Forlenza GP, Gallen G, Garg SK, Gershenoff DC, Gonder-Frederick LA, Haidar A, Hartnell S, Heinemann L, Heller S, Hirsch IB, Hood KK, Isaacs D, Klonoff DC, Kordonouri O, Kowalski A, Laffel L, Lawton J, Lal RA, Leelarathna L, Maahs DM, Murphy HR, Norgaard K, O'Neal D, Oser S, Oser T, Renard E, Riddell MC, Rodbard D, Russell SJ, Schatz DA, Shah VN, Sherr JL, Simonson GD, Wadwa RP, Ward C, Weinzimer SA, Wilmot EG, Battelino T. Consensus Recommendations for the Use of Automated Insulin Delivery Technologies in Clinical Practice. Endocr Rev. 2023 Mar 4;44(2):254-280. doi: 10.1210/endrev/bnac022. PMID 36066457
- [Background] Guerci B, Sauvanet JP. Subcutaneous insulin: pharmacokinetic variability and glycemic variability. Diabetes Metab. 2005 Sep;31(4 Pt 2):4S7-4S24. doi: 10.1016/s1262-3636(05)88263-1. PMID 16389894
- [Background] McAuley SA, Horsburgh JC, Ward GM, La Gerche A, Gooley JL, Jenkins AJ, MacIsaac RJ, O'Neal DN. Insulin pump basal adjustment for exercise in type 1 diabetes: a randomised crossover study. Diabetologia. 2016 Aug;59(8):1636-44. doi: 10.1007/s00125-016-3981-9. Epub 2016 May 11. PMID 27168135
- [Background] Paldus B, Morrison D, Zaharieva DP, Lee MH, Jones H, Obeyesekere V, Lu J, Vogrin S, La Gerche A, McAuley SA, MacIsaac RJ, Jenkins AJ, Ward GM, Colman P, Smart CEM, Seckold R, King BR, Riddell MC, O'Neal DN. A Randomized Crossover Trial Comparing Glucose Control During Moderate-Intensity, High-Intensity, and Resistance Exercise With Hybrid Closed-Loop Insulin Delivery While Profiling Potential Additional Signals in Adults With Type 1 Diabetes. Diabetes Care. 2022 Jan 1;45(1):194-203. doi: 10.2337/dc21-1593. PMID 34789504
- [Background] Mallad A, Hinshaw L, Schiavon M, Dalla Man C, Dadlani V, Basu R, Lingineni R, Cobelli C, Johnson ML, Carter R, Kudva YC, Basu A. Exercise effects on postprandial glucose metabolism in type 1 diabetes: a triple-tracer approach. Am J Physiol Endocrinol Metab. 2015 Jun 15;308(12):E1106-15. doi: 10.1152/ajpendo.00014.2015. Epub 2015 Apr 21. PMID 25898950
- [Background] Buehler LA, Noe D, Knapp S, Isaacs D, Pantalone KM. Ketogenic diets in the management of type 1 diabetes: Safe or safety concern? Cleve Clin J Med. 2021 Oct 1;88(10):547-555. doi: 10.3949/ccjm.88a.20121. PMID 34598919
- [Background] Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Research Group; Nathan DM, Zinman B, Cleary PA, Backlund JY, Genuth S, Miller R, Orchard TJ. Modern-day clinical course of type 1 diabetes mellitus after 30 years' duration: the diabetes control and complications trial/epidemiology of diabetes interventions and complications and Pittsburgh epidemiology of diabetes complications experience (1983-2005). Arch Intern Med. 2009 Jul 27;169(14):1307-16. doi: 10.1001/archinternmed.2009.193. PMID 19636033
- [Background] Weight gain associated with intensive therapy in the diabetes control and complications trial. The DCCT Research Group. Diabetes Care. 1988 Jul-Aug;11(7):567-73. doi: 10.2337/diacare.11.7.567. PMID 2904881
- [Background] Russo G, De Cosmo S, Di Bartolo P, Lucisano G, Manicardi V, Nicolucci A, Rocca A, Rossi MC, Di Cianni G, Candido R; AMD Annals Study Group. The quality of care in type 1 and type 2 diabetes - A 2023 update of the AMD Annals initiative. Diabetes Res Clin Pract. 2024 Jul;213:111743. doi: 10.1016/j.diabres.2024.111743. Epub 2024 Jun 13. PMID 38878867
- [Background] Musil F, Smahelova A, Blaha V, Hyspler R, Ticha A, Lesna J, Zadak Z, Sobotka L. Effect of low calorie diet and controlled fasting on insulin sensitivity and glucose metabolism in obese patients with type 1 diabetes mellitus. Physiol Res. 2013;62(3):267-76. doi: 10.33549/physiolres.932381. Epub 2013 Mar 14. PMID 23489182
- [Background] Barrea L, Caprio M, Camajani E, Verde L, Perrini S, Cignarelli A, Prodam F, Gambineri A, Isidori AM, Colao A, Giorgino F, Aimaretti G, Muscogiuri G. Ketogenic nutritional therapy (KeNuT)-a multi-step dietary model with meal replacements for the management of obesity and its related metabolic disorders: a consensus statement from the working group of the Club of the Italian Society of Endocrinology (SIE)-diet therapies in endocrinology and metabolism. J Endocrinol Invest. 2024 Mar;47(3):487-500. doi: 10.1007/s40618-023-02258-2. Epub 2024 Jan 18. PMID 38238506
- [Background] Gardemann C, Knowles S, Marquardt T. Managing type 1 diabetes mellitus with a ketogenic diet. Endocrinol Diabetes Metab Case Rep. 2023 Aug 16;2023(3):23-0008. doi: 10.1530/EDM-23-0008. Print 2023 Aug 1. PMID 37584373
- [Background] Corbin KD, Driscoll KA, Pratley RE, Smith SR, Maahs DM, Mayer-Davis EJ; Advancing Care for Type 1 Diabetes and Obesity Network (ACT1ON). Obesity in Type 1 Diabetes: Pathophysiology, Clinical Impact, and Mechanisms. Endocr Rev. 2018 Oct 1;39(5):629-663. doi: 10.1210/er.2017-00191. PMID 30060120
- [Background] Fang M, Jeon Y, Echouffo-Tcheugui JB, Selvin E. Prevalence and Management of Obesity in U.S. Adults With Type 1 Diabetes. Ann Intern Med. 2023 Mar;176(3):427-429. doi: 10.7326/M22-3078. Epub 2023 Feb 14. No abstract available. PMID 36780652
- [Background] Foster NC, Beck RW, Miller KM, Clements MA, Rickels MR, DiMeglio LA, Maahs DM, Tamborlane WV, Bergenstal R, Smith E, Olson BA, Garg SK. State of Type 1 Diabetes Management and Outcomes from the T1D Exchange in 2016-2018. Diabetes Technol Ther. 2019 Feb;21(2):66-72. doi: 10.1089/dia.2018.0384. Epub 2019 Jan 18. PMID 30657336